CLINICAL TRIAL: NCT05750290
Title: CKD-702 Plus Irinotecan as a ≥3L Therapy for Gastric and Gastroesophageal Junction Adenocarcinomas Overexpressing EGFR or MET
Brief Title: CKD-702 Plus Irinotecan in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100945
Record Dates: First submitted 2023-02-09; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CKD-702 in combination with irinotecan (Experimental)
  Interventions: Drug: CKD-702 in combination with irinotecan

INTERVENTIONS:
Drug: CKD-702 in combination with irinotecan — CKD-702 and irinotecan will be intravenously administered every 2 weeks.

SUMMARY:
CKD-702 is a tetravalent bispecific IgG1 targeting hepatocyte growth factor receptor (MET) and epidermal growth factor receptor (EGFR). The investigators will test a hypothesis that CKD-702 may augment the efficacy of biweekly irinotecan as a 3L or later therapy for gastric cancer overexpressing either MET or EGFR.

ELIGIBILITY:
Inclusion Criteria:

* Failed 2 or more lines of chemotherapy
* Tumor overexpressing either MET or EGFR
* Measurable lesion

Exclusion Criteria:

* Prior treatment with anti-MET/EGFR bispecific antibody

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Best objective response rate | Through study completion, an average of 24 weeks
  RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No